CLINICAL TRIAL: NCT07319169
Title: The Value of Spleen Stiffness Measurement in Patients With PBC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VasMe PBC
Record Dates: First submitted 2025-12-05; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-11

CONDITIONS: Primary Biliary Cholangitis; Spleen Stiffness
Keywords: spleen stiffness; primary biliairy cholangitis
MeSH Terms: conditions — Liver Cirrhosis, Biliary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Spleen stiffness measurement (Experimental)
  Interventions: Procedure: Spleen stiffness measurement

INTERVENTIONS:
Procedure: Spleen stiffness measurement — spleen stiffness measurement - during FibroScan

SUMMARY:
Recent evidence suggests that combining liver stiffness measurement (LSM) with spleen stiffness measurement (SSM) significantly improves risk stratification in patients with PBC. In a study the addition of spleen stiffness to liver stiffness enhanced the prediction of liver decompensation, providing a more precise evaluation of portal hypertension. Furthermore, when combined with platelet count, this approach effectively identified patients with a low probability of harboring HRVs. This could allow clinicians to safely avoid unnecessary endoscopic procedures in selected patients, improving patient comfort and reducing healthcare costs. Therefore, our patients participating in this trial will undergo follow up (every 6 months) as per Standard of care. This includes a blood draw, FibroScan and Ultrasound. Together with this, 2 questionnaires will be completed (not as per SOC) and during the FibroScan, a spleen stiffness measurement will be performed.

ELIGIBILITY:
Inclusion Criteria:

* ≥18y
* Out-patient, followed at the UZ Brussels
* Diagnosis of PBC based on cholestasis, AMA positivity and/or biopsy.
* Under treatment with ursodeoxycholic acid and/or bezafibrate

Exclusion Criteria:

* <18y
* Contra-indication for transient elastography (Fibroscan®) such as ascites or overt heart failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Correlation between spleen stiffness measurement and biochemical assessment of severity of PBC. | from signing the ICF till end of study (could be up to 5 years, assessments are done every 6 months)
Correlation between spleen stiffness measurement and clinical signs of portal hypertension, liver related events and PH-related bleeding | from signing the ICF till end of study (could be up to 5 years, assessments are done every 6 months)
Correlation between spleen stiffness measurement and endoscopic signs of portal hypertension, liver related events and PH-related bleeding | from signing the ICF till end of study (could be up to 5 years, assessments are done every 6 months)
Correlation between spleen stiffness measurement and quality of life assessment of severity of PBC. | from signing the ICF till end of study (could be up to 5 years, assessments are done every 6 months)
Evaluation of the evolution of liver or spleen stiffness on treatment of PBC | from signing the ICF till end of study (could be up to 5 years, assessments are done every 6 months)
  liver or spleen stiffness measurement is done using FibroScan

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No